CLINICAL TRIAL: NCT02116192
Title: Early Intervention and Prevention of Non-Alcoholic Fatty Liver Disease in Adolescents
Acronym: NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K12HD055894 (NIH)
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Non-alcoholic Fatty Liver Disease; Adolescent
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- General Healthy Diet (Active Comparator): Control: General Healthy Diet (Prescribed Hypocaloric regimen to promote 7% initial weight loss via 25-30kCal/kg; 50-60% CHO, 15-20% Protein, 20-30% Fat)
  Interventions: Behavioral: General Healthy Diet
- Low-fructose, reduced carbohydrate diet (Experimental): Intervention: Low Carbohydrate (Low Fructose and Sucrose) Diet (Prescribed Hypocaloric regimen to promote 7% initial weight loss via 25-30kCal/kg;40-45% CHO, 20-25% Protein, 30-40% Fat)
  ● Aim for less than 25g fructose daily.
  Interventions: Behavioral: Experimental: Low-fructose, reduced carbohydrate diet

INTERVENTIONS:
Behavioral: Experimental: Low-fructose, reduced carbohydrate diet — Low Carbohydrate (Low Fructose and Sucrose) Diet (Prescribed Hypocaloric regimen to promote 7% initial weight loss via 25-30kCal/kg;40-45% CHO, 20-25% Protein, 30-40% Fat)
  ● Aim for less than 25g fructose daily.
  Arms: Low-fructose, reduced carbohydrate diet
Behavioral: General Healthy Diet — Prescribed Hypocaloric regimen to promote 7% initial weight loss via 25-30kCal/kg; 50-60% CHO, 15-20% Protein, 20-30% Fat
  Arms: General Healthy Diet

SUMMARY:
This research study intends to learn about whether early intervention can help to prevent non-alcoholic fatty liver disease (NAFLD) in adolescents. Potentially eligible adolescents who are seen at the University of Wisconsin (UW) Pediatric Fitness Clinic will be asked to join the study. Patients who agree to participate in the study will be randomized into either the intervention group or the control group. The intervention group will follow a low-fructose diet. In addition, participants will be asked to return to the clinic for 4 follow-up visits during a 6-month interval.

DETAILED DESCRIPTION:
This will be a prospective, randomized, controlled trial for obese adolescents. Sixty obese youth (male and female), age 11-17 years with BMI >95 %tile for age and sex and one parent/guardian will be recruited for inclusion into the study at an initial pediatric fitness clinic visit. Consented subjects will be stratified by gender and ethnicity and randomized into low fructose or standard weight loss dietary intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* 11-17 years of age
* BMI >95%tile for age and sex
* Being seen for an initial clinic visit at the UW Pediatric Fitness Clinic
* Parent willing to participate in study

Exclusion Criteria:

* History of chronic disease that effects hepatic or renal function including: Type 1 or Type 2 diabetes mellitus, known liver disease or other chronic illness.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Hepatic triglyceride content measured by Magnetic resonance (MR) PDFF | 6 months

SECONDARY OUTCOMES:
Metabolic biomarkers | 6 months
  Including waist circumference (WC), blood pressure (BP), insulin resistance measured by homeostasis model assessment (HOMA-IR), lipids, ALT, androgens, and visceral and subcutaneous adiposity (by MR PDFF), and cardiovascular fitness (sub-maxVO2 test), in low carbohydrate/low fructose and standard weight-reduction diet groups
PNPLA3 genotype | 6 months
Novel free breathing hepatic MR PDFF protocol | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Rehm, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Research Park Clinic, Madison, Wisconsin, United States

REFERENCES:
- [Background] American Gastroenterological Association. American Gastroenterological Association medical position statement: nonalcoholic fatty liver disease. Gastroenterology. 2002 Nov;123(5):1702-4. doi: 10.1053/gast.2002.36569. No abstract available. PMID 12404244
- [Background] Assy N, Nasser G, Kamayse I, Nseir W, Beniashvili Z, Djibre A, Grosovski M. Soft drink consumption linked with fatty liver in the absence of traditional risk factors. Can J Gastroenterol. 2008 Oct;22(10):811-6. doi: 10.1155/2008/810961. PMID 18925303
- [Background] Brunt EM. Nonalcoholic steatohepatitis. Semin Liver Dis. 2004 Feb;24(1):3-20. doi: 10.1055/s-2004-823098. PMID 15085483
- [Background] Brunt EM. Pathology of nonalcoholic steatohepatitis. Hepatol Res. 2005 Oct;33(2):68-71. doi: 10.1016/j.hepres.2005.09.006. Epub 2005 Oct 7. PMID 16214395
- [Background] Chitturi S, Farrell GC. Etiopathogenesis of nonalcoholic steatohepatitis. Semin Liver Dis. 2001;21(1):27-41. doi: 10.1055/s-2001-12927. PMID 11296694
- [Background] Clark JM. The epidemiology of nonalcoholic fatty liver disease in adults. J Clin Gastroenterol. 2006 Mar;40 Suppl 1:S5-10. doi: 10.1097/01.mcg.0000168638.84840.ff. PMID 16540768
- [Background] Curtis VA, Carrel AL, Eickhoff JC, Allen DB. Gender and race influence metabolic benefits of fitness in children: a cross-sectional study. Int J Pediatr Endocrinol. 2012 Mar 15;2012(1):4. doi: 10.1186/1687-9856-2012-4. PMID 22420715
- [Background] Della Corte C, Alisi A, Saccari A, De Vito R, Vania A, Nobili V. Nonalcoholic fatty liver in children and adolescents: an overview. J Adolesc Health. 2012 Oct;51(4):305-12. doi: 10.1016/j.jadohealth.2012.01.010. Epub 2012 Mar 13. PMID 22999829
- [Background] Denzer C, Thiere D, Muche R, Koenig W, Mayer H, Kratzer W, Wabitsch M. Gender-specific prevalences of fatty liver in obese children and adolescents: roles of body fat distribution, sex steroids, and insulin resistance. J Clin Endocrinol Metab. 2009 Oct;94(10):3872-81. doi: 10.1210/jc.2009-1125. Epub 2009 Sep 22. PMID 19773396
- [Background] Dishman RK, Dunn AL, Sallis JF, Vandenberg RJ, Pratt CA. Social-cognitive correlates of physical activity in a multi-ethnic cohort of middle-school girls: two-year prospective study. J Pediatr Psychol. 2010 Mar;35(2):188-98. doi: 10.1093/jpepsy/jsp042. Epub 2009 May 25. PMID 19468040
- [Background] Dunn W, Schwimmer JB. The obesity epidemic and nonalcoholic fatty liver disease in children. Curr Gastroenterol Rep. 2008 Feb;10(1):67-72. doi: 10.1007/s11894-008-0011-1. PMID 18417045
- [Background] Feldstein AE, Charatcharoenwitthaya P, Treeprasertsuk S, Benson JT, Enders FB, Angulo P. The natural history of non-alcoholic fatty liver disease in children: a follow-up study for up to 20 years. Gut. 2009 Nov;58(11):1538-44. doi: 10.1136/gut.2008.171280. Epub 2009 Jul 21. PMID 19625277
- [Background] Kawasaki T, Igarashi K, Koeda T, Sugimoto K, Nakagawa K, Hayashi S, Yamaji R, Inui H, Fukusato T, Yamanouchi T. Rats fed fructose-enriched diets have characteristics of nonalcoholic hepatic steatosis. J Nutr. 2009 Nov;139(11):2067-71. doi: 10.3945/jn.109.105858. Epub 2009 Sep 23. PMID 19776184
- [Background] Loomba R, Sirlin CB, Schwimmer JB, Lavine JE. Advances in pediatric nonalcoholic fatty liver disease. Hepatology. 2009 Oct;50(4):1282-93. doi: 10.1002/hep.23119. PMID 19637286
- [Background] Ludwig J, Viggiano TR, McGill DB, Oh BJ. Nonalcoholic steatohepatitis: Mayo Clinic experiences with a hitherto unnamed disease. Mayo Clin Proc. 1980 Jul;55(7):434-8. PMID 7382552
- [Background] Lytle LA, Murray DM, Evenson KR, Moody J, Pratt CA, Metcalfe L, Parra-Medina D. Mediators affecting girls' levels of physical activity outside of school: findings from the trial of activity in adolescent girls. Ann Behav Med. 2009 Oct;38(2):124-36. doi: 10.1007/s12160-009-9127-2. Epub 2009 Dec 12. PMID 20012810
- [Background] McCullough AJ. The clinical features, diagnosis and natural history of nonalcoholic fatty liver disease. Clin Liver Dis. 2004 Aug;8(3):521-33, viii. doi: 10.1016/j.cld.2004.04.004. PMID 15331061
- [Background] Miller WR. What really drives change? Addiction. 1993 Nov;88(11):1479-80. doi: 10.1111/j.1360-0443.1993.tb03133.x. No abstract available. PMID 8286993
- [Background] Nomura K, Yamanouchi T. The role of fructose-enriched diets in mechanisms of nonalcoholic fatty liver disease. J Nutr Biochem. 2012 Mar;23(3):203-8. doi: 10.1016/j.jnutbio.2011.09.006. Epub 2011 Nov 29. PMID 22129639
- [Background] Park YK, Yetley EA. Intakes and food sources of fructose in the United States. Am J Clin Nutr. 1993 Nov;58(5 Suppl):737S-747S. doi: 10.1093/ajcn/58.5.737S. PMID 8213605
- [Background] Pozzato C, Verduci E, Scaglioni S, Radaelli G, Salvioni M, Rovere A, Cornalba G, Riva E, Giovannini M. Liver fat change in obese children after a 1-year nutrition-behavior intervention. J Pediatr Gastroenterol Nutr. 2010 Sep;51(3):331-5. doi: 10.1097/MPG.0b013e3181d70468. PMID 20562718
- [Background] Sallis JF, McKenzie TL, Conway TL, Elder JP, Prochaska JJ, Brown M, Zive MM, Marshall SJ, Alcaraz JE. Environmental interventions for eating and physical activity: a randomized controlled trial in middle schools. Am J Prev Med. 2003 Apr;24(3):209-17. doi: 10.1016/s0749-3797(02)00646-3. PMID 12657338
- [Background] Schwimmer JB. Definitive diagnosis and assessment of risk for nonalcoholic fatty liver disease in children and adolescents. Semin Liver Dis. 2007 Aug;27(3):312-8. doi: 10.1055/s-2007-985075. PMID 17682977
- [Background] Szczepaniak LS, Nurenberg P, Leonard D, Browning JD, Reingold JS, Grundy S, Hobbs HH, Dobbins RL. Magnetic resonance spectroscopy to measure hepatic triglyceride content: prevalence of hepatic steatosis in the general population. Am J Physiol Endocrinol Metab. 2005 Feb;288(2):E462-8. doi: 10.1152/ajpendo.00064.2004. Epub 2004 Aug 31. PMID 15339742
- [Background] Williams KH, Shackel NA, Gorrell MD, McLennan SV, Twigg SM. Diabetes and nonalcoholic Fatty liver disease: a pathogenic duo. Endocr Rev. 2013 Feb;34(1):84-129. doi: 10.1210/er.2012-1009. Epub 2012 Dec 13. PMID 23238855